CLINICAL TRIAL: NCT03319511
Title: Comparison Between Thoracic Para-vertebral Block and Segmental Thoracic Spinal Anesthesia in Breast Cancer Surgery
Brief Title: Thoracic Spinal Anesthesia in Awake Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alaa Mazy (Other)
Responsible Party: Sponsor-Investigator, Alaa Mazy, Associate professor of anesthesia and surgical intensive care, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD/15.05.91
Record Dates: First submitted 2017-10-16; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: thoracic spinal; awake mastectomy; paravertebral block; analgesia; ultrasound; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: a dorsal thoracic gauze cover.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paravertebral group (Active Comparator): ultrasound guided, in sitting position, or lateral position, at T2 and T4 levels, using 22 G spinal needle, in plane technique, traversing the costo-transverse ligament
  Interventions: Other: paravertebral group
- spinal group (Experimental): Ultrasound guided, In the lateral decubitus or sitting position, the puncture performed via para-median approach, at the T4-T5 or T5-T6 interspace, with a 27G spinal needle. After piercing the ligamentum flavum, the needle's stylet removed and the hub observed for free flow of CSF; injection when there is a flow of clear CSF.
  Interventions: Other: spinal group

INTERVENTIONS:
Other: spinal group — plain bupivacaine 0.5%,1.5 ml plus dexmedetomidine 5 μg. once injection.
  Other Names: STSB
  Arms: spinal group
Other: paravertebral group — plain bupivacaine 0.5%, 0.3 ml (1.5 mg)/kg plus dexmedetomidine 0.5 μg /kg divided between the T2 and T4 levels.
  Other Names: TPVB
  Arms: paravertebral group

SUMMARY:
General anesthesia is the conventional technique used for breast surgery. breast surgery is associated with a high incidence of postoperative pain, it is estimated that over 50 % of women suffer chronic pain following breast cancer surgery. Regional anesthesia is a good alternative to general anesthesia for breast cancer surgery, providing superior analgesia and fewer side effects related to a standard opiate-based analgesia. there is no evident optimal regional techniques for operative procedures on the breast and axilla, like high thoracic epidural, cervical epidural, paravertebral block, intrerpleural block, PECs block, serratus plane block and segmental thoracic spinal anesthesia. Regional anesthesia decreases operative stress, provides beneficial hemodynamic effects especially for critically ill patients and decreases postoperative morbidity and mortality. Also it reduces post-operative nausea and vomiting and provides prolonged post-operative sensory block, minimizing narcotic requirements. Additionally, this application positively affects the early start of feeding and mobilization.

DETAILED DESCRIPTION:
Thoracic paravertebral block (TPVB) is an alternative method to general anesthesia for patients undergoing breast surgery, because it provides a safe anesthesia with balanced hemodynamic response with unilateral somatic and sympathetic blockade, allows postoperative analgesia lowering narcotic usage , minimal nausea and vomiting rate, early discharge and low cost.

Segmental thoracic spinal anesthesia have introduced for cardiac surgery in adults and children in the early 1990's. Kowalewski et al., performed over 10000 cases of spinal injections without a single case of spinal/epidural hematoma or any neurological complications, also segmental thoracic spinal anesthesia has been used successfully for laparoscopic cholecystectomy and abdominal surgeries. It has some advantages when compared with general anesthesia and can be a sole anesthetic in breast cancer surgery with axillary lymph node clearance especially in critical cases. Among its advantages are the quality of postoperative analgesia, lower incidence of nausea and vomiting, and shorter recovery time, with the consequent early hospital discharge. The dose of the anesthetic is exceedingly low, compared with lumbar spinal anesthesia, given the highly specific block to only certain nerve functions along a section of the cord, there is no blockade of the lower extremities. This means that a significantly larger portion of the body experiences no venal dilation, and may offer a compensatory buffer to adverse changes in blood pressure intra-operatively. there was no recorded of neurological complications.The incidence of parasthesia in a study with 300 patients subjected to thoracic spinal puncture at T10-11 was 4.67% in the cut needle group and 8.67% in the pencil point needle group, similar to that reported in lumbar spinal anesthesia.The aim of the present study is the comparison between two sole regional anesthetic techniques, thoracic para-vertebral block and segmental thoracic spinal anesthesia in breast cancer surgery especially for critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

ASA II, III, IV patients may have:

1. Cardiovascular disease (e.g., rheumatic heart, systemic hypertension, ischemic heart)
2. Lung disease (e.g., bronchial asthma, COPD)
3. Renal disease (e.g., renal failure, polycystic kidney)
4. Liver disease (e.g., cirrhosis, hepatitis)
5. Endocrine disease (e.g., diabetes mellitus)

Exclusion Criteria:

1. Patient refusal
2. Contraindication to regional anesthesia (coagulopathy, local infection),
3. Spinal deformities.
4. An allergy to α 2 adrenergic agonist local anesthetic drugs.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients scheduled for unilateral modified radical mastectomy with axillary dissection for breast cancer.
Enrollment: 70 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2016-11-12 (Actual); Study Completion 2016-11-12 (Actual)

PRIMARY OUTCOMES:
the block success rate. | within 30 min of injection
  in number, defined as complete sensory block in all dermatomes (T1-T6 ).

SECONDARY OUTCOMES:
The paravertebral onset of sensory block | 5, 10, 15, 20, 52, 30 minutes after injection.
  tested for loss of sensation, with a needle along the anterior axillary line from T1-T6 on the blocked side.
The spinal onset of sensory block | 2, 4, 6, 8, 10, 12, 14 minutes after injection.
  tested for loss of sensation, with a needle along the anterior axillary line from T1-T6 on the blocked side.
The power of hand grip (T1/ C8) | 5, 10, 15, 20, 52, 30 minutes after injection.
  four grades (0-3), 0= no motor block, 1= partial, 2= almost complete, 3= complete motor block.
The power of wrist flexion (C8/C7) | 5, 10, 15, 20, 52, 30 minutes after injection.
  four grades (0-3), 0= no motor block, 1= partial, 2= almost complete, 3= complete motor block.
The power of elbow flexion (C6/ C5) | 5, 10, 15, 20, 52, 30 minutes after injection.
  four grades (0-3), 0= no motor block, 1= partial, 2= almost complete, 3= complete motor block.
The onset time of lower limb motor block (Bromage 3) | 5, 10, 15, 20, 25, 30 minutes after injection.
  in minutes, 3= unable to move legs or feet.
The duration of lower limb motor block (Bromage 0) | 30, 45, 60, 90,120, 150 minutes after injection.
  minutes, 0= free movement of legs and feet
Ramsey sedation scale | 0 (basal), then1, 5, 10, 15, 30, 45, 60, 75, 90, 120 minutes from injection time, then 1, 4, 5, 6, 7, 8, 12, 18, 24 hours starting after the end of operation.
  (1 = awake, conscious, no sedation; 2 = calm and compose; 3 = awake on verbal command; 4 = brisk response to gentle tactile stimulation; 5 = awake on vigorous shaking; 6 = unarousable).
Heart rate | 0= basal, then 1, 5, 10, 15, 30, 45, 60, 75, 90, 120 minutes from injection time, then 1, 4, 5, 6, 7, 8, 12, 18, 24 hours starting after the end of operation.
  beat/minute
Systolic blood pressure | 0= basal, then 1, 5, 10, 15, 30, 45, 60, 75, 90, 120 minutes from injection time, then 1, 4, 5, 6, 7, 8, 12, 18, 24 hours starting after the end of operation.
  millimeter mercury
Mean blood pressure | 0= basal, then 1, 5, 10, 15, 30, 45, 60, 75, 90, 120 minutes from injection time, then 1, 4, 5, 6, 7, 8, 12, 18, 24 hours starting after the end of operation.
  millimeter mercury
Total ephedrine consumption | intraoperative
  milligram, Hypotension defined as 20% drop in baseline blood pressure or systolic pressure below 90 mm Hg)
Total atropine consumption | intraoperative
  milligram, Bradycardia defined as heart rate below 50 beat/minute
Total Midazolam consumption | intraoperative
  milligram,
Hypotension episodes | Intraoperative and postoperative for 24 hours.
  in number. Hypotension (20% drop in baseline blood pressure or systolic pressure below 90 mm Hg).
Bradycardia episodes | Intraoperative and postoperative for 24 hours.
  In number. Bradycardia defined as heart rate below 50 beat/minute
Hypoxia episodes | Intraoperative and postoperative for 24 hours.
  In number. Hypoxia is defined as defined as respiratory rate <10 breath/ minutes or oxygen saturation less than 90%.
incidence of nausea | Intraoperative and postoperative for 24 hours.
  In number.
incidence of vomiting | Intraoperative and postoperative for 24 hours.
  In number.
the incidence of pneumothorax. | intraoperative and postoperative for 6 hours.
  in numbers. confirmed by plane X-ray
The incidence of post-dural puncture headache. | postoperative for 72 hours.
  in numbers.
The duration of upper limb motor block, | 15, 30, 45, 60, 90 minutes after injection.
  minutes. starting from the time of score 3 to score 0 (0= no motor block).
Visual analog scale | at 0, 4, 5, 6, 7, 8, 12, 18, 24 hours postoperative.
  a 0-10 cm scale, 0 represents no pain and 10 is the worst pain.
The total mepridine consumption. | postoperative for 24 hours.
  milligram
satisfaction of the patient | after 24 hours from the end of operation.
  scale from 0-10, 10= the highest.
satisfaction of the surgeon | within 2 hours from the end of operation.
  scale from 0-10, 10= the highest.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncolgy Center, Mansoura University,, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: after publication, for no limit
Access Criteria: e mail: alaa_mazy@yahoo.com